CLINICAL TRIAL: NCT06799637
Title: A Phase 1, Open-Label, Multicenter Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Antitumor Efficacy of XNW28012 in Subjects with Advanced Solid Tumors
Brief Title: Study of XNW28012 in Subjects with Advanced Solid Tumors Who Failed Standard Treatments
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Evopoint Biosciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XNW28012-I/II-01
Record Dates: First submitted 2024-12-25; First posted 2025-01-29 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2024-12

CONDITIONS: Advanced Solid Tumors; Pancreatic Carcinoma; Ovarian Cancer; Cervical Cancers
Keywords: XNW28012
MeSH Terms: conditions — Pancreatic Neoplasms; Ovarian Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Bayesian Optimal Interval (BOIN) method will be used for the dose escalation part. (Other): Based on the toxicology data from preclinical studies, the Bayesian Optimal Interval (BOIN) method will be used for the dose escalation part with preset doses at 0.6 mg/kg, 1.2 mg/kg, 2.4 mg/kg, 3.6 mg/kg, 4.8 mg/kg, 6.0 mg/kg, and 7.5 mg/kg. Eligible subjects will receive XNW28012 every 3 weeks (Q3W) until intolerant toxicity, progression of disease with no clinical benefit, or withdrawal of informed consent. The first treatment cycle will be the dose limiting toxicity (DLT) assessment period. The safety, tolerability, and occurrence of DLTs will be assessed during the DLT period. The proposed dose escalation plan is shown below.
  Interventions: Drug: XNW28012

INTERVENTIONS:
Drug: XNW28012 — Eligible subjects will receive XNW28012 every 3 weeks (Q3W) until intolerant toxicity, progression of disease with no clinical benefit, or withdrawal of informed consent.

SUMMARY:
This is an open-label, dose escalation, multicenter, phase 1, first-in-human study of XNW28012 in subjects with advanced solid tumors who have failed current standard anti-tumor therapies or are intolerant to such therapies. The study consists of two parts: a dose escalation part and a dose expansion part.

ELIGIBILITY:
Inclusion Criteria:

1. For the dose escalation part: subjects with histologically or cytologically confirmed advanced and/or metastatic solid tumors who have failed the established standard anti-cancer therapies for a given tumor type or have been intolerant to such therapies.
2. For the dose expansion part: subjects must have a histological or cytological diagnosis of progressive, locally advanced, and/or metastatic ovarian cancer, cervical cancer, pancreatic cancer, or colorectal cancer (CRC) who have failed the following anti-cancer therapies: Ovarian cancer, Cervical cancer, Pancreatic cancer, Colorectal cancer.
3. Age ≥ 18 years old at the time of consent.
4. Subjects must have at least 1 measurable lesion as defined per RECIST version 1.1 (for dose expansion part only).
5. Subjects must have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale. ECOG status of 2 can be allowed if it is a result of disease progression and warrants discussion with the medical monitor.
6. Subjects must have adequate organ function within 7 days prior to the first study drug administration, as indicated by the flaboratory values:
7. Life expectancy of at least 12 weeks.
8. Females of childbearing potential must have a negative pregnancy test within 7 days prior to the first dose of study drug. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
9. Non-sterile subjects must be willing to use a highly effective contraception (e.g., IUD, pill, or condom) for the duration of the study and for 6 months after the last dose of study drug unless their partner is sterilized.
10. Subjects are able to provide written informed consent, understand and are willing to comply with the requirements of the study.

Exclusion Criteria:

1. A history of severe infusion reactions to other monoclonal antibodies/antibody drug conjugates (ADCs) or allergic reactions to any components of XNW28012.
2. Any anti-tumor therapy within 28 days prior to the first dose, including but not limited to: small molecules, immunotherapy, chemotherapy, monoclonal antibodies, or any other experimental drugs.
3. Any active malignancy, with the exception of the specific types of cancers under investigation in this study and any locally recurring cancer that has been treated curatively .
4. Have received a live vaccine within 4 weeks prior to the first dose of study drug. Note: Seasonal vaccines for influenza are generally inactivated vaccines and are allowed; however, intranasal influenza vaccines will not be allowed if they are attenuated live vaccines.
5. Have received granulocyte colony stimulating factor (G-CSF) or granulocyte / macrophage colony stimulating factor support within 1 week before screening, or pegylated G-CSF within 2 weeks before screening.
6. Subjects with toxicities (as a result of prior anti-cancer therapy) which have not improved to CTCAE grade ≤1 or stabilized, except those AEs not considered as a likely safety risk (e.g., alopecia).
7. Any history of intracerebral arteriovenous malformation, cerebral aneurysm, or stroke (transient ischemic attack) ≤ 3 months prior to screening is allowed if stable.
8. Any of the hematological risk factors:
9. Subjects who are unwilling or unable to provide tumor tissue samples that meet the requirements for tissue factor (TF) expression testing.

11. Clinically significant cardiovascular/cerebrovascular conditions. 12. Active ocular surface disease at screening, or subjects with any prior episode of cicatricial conjunctivitis.

13. Any history of Toxic Epidermal Necrolysis (TEN) or Steven Johnson Syndrome. 14. Subjects who have undergone major surgery within 28 days prior to the first dose of study drug, except if the procedure is minimally invasive (for example, introduction of peripherally inserted central catheter [PICC] line).

and so on.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Ph 1: Incidence and severity of treatment-emergent adverse events (AEs) [Safety and Tolerability]. | through study completion, an average of 1 year
  Incidence and severity of adverse events that are graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) version 5.0.
Ph 2: To evaluate the antitumor efficacy of XNW28012 at the recommended Part 2 dose. | through study completion, an average of 1 year
  ORR per RECIST1.1 assessed by Investigators.

SECONDARY OUTCOMES:
Ph 1:Maximum tolerated dose (MTD) and/or the recommended Part 2 dose. | The first 21-day cycle of therapy
  To determine the maximum tolerated dose (MTD) and the recommended Part 2 dose with XNW28012;
Ph 1/II: Maximum (peak) observed concentration (Cmax) of XNW28012. | through study completion, an average of 1 year
  Blood samples were collected at specified intervals for the determination of Cmax.
Ph 1/II: Maximum (peak) observed concentration (Cmax) of total antibody of XNW28012.. | through study completion, an average of 1 year
  Blood samples were collected at specified intervals for the determination of Cmax.
Ph 1/II: Maximum (peak) observed concentration (Cmax) of YL0010014 | through study completion, an average of 1 year
  Blood samples were collected at specified intervals for the determination of Cmax.
Ph 1/II: Anti-drug antibody (ADA) | through study completion, an average of 1 year
  To assess the incidence of anti-drug antibody (ADA) against XNW28012
Ph I/II：Objective response rate (ORR) | Efficacy assessments will be performed at screening (≤ 28 days prior to the first dose), every 6 weeks for 24 weeks after the first dose, and every 12 weeks after the 24 weeks response assessments until disease progression (up to 1 year).
  ORR is defined as the proportion of subjects who have a confirmed CR or a PR per RECIST 1.1 assessed by Investigator.
Ph I/II: Disease control rate (DCR) | Efficacy assessments will be performed at screening (≤ 28 days prior to the first dose), every 6 weeks for 24 weeks after the first dose, and every 12 weeks after the 24 weeks response assessments until disease progression (up to 1 year).
  Rate of complete response [CR], partial response [PR], and stable disease per RECIST1.1 assessed by Investigator.
Ph I/II：Progression free survival (PFS) | Efficacy assessments will be performed at screening (≤ 28 days prior to the first dose), every 6 weeks for 24 weeks after the first dose, and every 12 weeks after the 24 weeks response assessments until disease progression (up to 1 year).
  Progression free survival (PFS) per RECIST1.1 assessed by Investigator
Ph I/II: Duration of response (DOR) | Efficacy assessments will be performed at screening (≤ 28 days prior to the first dose), every 6 weeks for 24 weeks after the first dose, and every 12 weeks after the 24 weeks response assessments until disease progression (up to 1 year).
  Duration of response (DOR) per RECIST1.1 assessed by Investigator.

OTHER OUTCOMES:
Ph 1/2: Tissue factor expression | At screening
  Correlation between tissue factor expression and the antitumor efficacy of XNW28012.

CONTACTS AND LOCATIONS:
Locations (24):
- China (24):
  - Second Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - The First Affiliated Hospital of University of Science and Technology of China, Hefei, Anhui
  - Beijing Friendship Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - Fujian Provincial Cancer Hospital, Fuzhou, Fujian
  - Sun Yat-sen Memorial Hospital, Sun Yat-sen University, Guangzhou, Guangdong
  - Affiliated Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - Affiliated Cancer Hospital of Harbin Medical University, Harbin, Heilongjiang
  - First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan
  - Hubei Cancer Hospital, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - The Second Xiangya Hospital Of Central South University, Changsha, Hunan
  - First Affiliated Hospital of Gannan Medical College, Ganzhou, Jiangxi
  - First Affiliated Hospital of Kunming Medical University, Yunnan, Kunming
  - Affiliated Hospital of Binzhou Medical College, Binzhou, Shandong
  - Jinan Central Hospital, Jinan, Shandong
  - Linyi Cancer Hospital, Linyi, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No